CLINICAL TRIAL: NCT02524899
Title: Guanfacine Enhancement of Working Memory: Prospects for Augmenting Cognitive Remediation in the Schizophrenia Spectrum
Brief Title: CRT-Guanfacine for SPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Margaret McNamara McClure, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 13-0109
Record Dates: First submitted 2015-08-10; First posted 2015-08-17 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Schizotypal Personality Disorder; SPD
Keywords: Schizotypal Personality Disorder; SPD; cognitive remediation therapy; CRT; guanfacine; cognitive impairment; working memory; pharmacological cognitive enhancing agent; neuropsychological testing; schizophrenia spectrum disorders; Personality Disorders
MeSH Terms: conditions — Schizotypal Personality Disorder; Cognitive Dysfunction; Personality Disorders | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Remediation Therapy and placebo (Active Comparator): 7.5 weeks of twice weekly cognitive remediation sessions
  Interventions: Behavioral: Cognitive Remediation Therapy; Drug: Placebo
- Guanfacine and CRT (Experimental): 7.5 weeks of twice weekly cognitive remediation sessions with 8 weeks of guanfacine
  Interventions: Behavioral: Cognitive Remediation Therapy; Drug: Guanfacine

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Cognitive Remediation Therapy (CRT) will consist of fifteen 45-minute, twice weekly sessions over 7.5 weeks. During each session, subjects, seated at a desk in a private interview room in our research office suite, will work through exercises that are part of the Psychological Software Services CogReHab program. The software to be used is a multimedia, Windows-based program that consists of exercises aimed at improving areas of deficit within the schizophrenia spectrum, such as executive function, working memory, and social cognition.
  Other Names: CRT
Drug: Guanfacine — After completing baseline cognitive testing, subjects will be randomized to guanfacine or placebo. Subjects in the active treatment arm will begin with a guanfacine dose of 0.5mg/day and be titrated up to a maximum of 2mg/day according to our well-tolerated protocol in schizophrenia subjects. The dosing schedule of active guanfacine will be as follows: 0.5mg/d for week 1, 1.0mg/d for week 2, 1.0 mg bid for weeks 3, 4, 5, 6, and 7 and 1.0mg/d for week 8.
  Arms: Guanfacine and CRT
Drug: Placebo — After completing baseline cognitive testing, subjects will be randomized to guanfacine or placebo. Subjects in placebo arm will have matching schedule as active arm.
  Arms: Cognitive Remediation Therapy and placebo

SUMMARY:
This is a study to assess the efficacy augmenting cognitive remediation therapy (CRT) with a pharmacological agent for individuals with schizotypal personality disorder (SPD). Impaired cognition, along with functional and social skill deficits, is a core feature of schizophrenia and schizophrenia spectrum disorders. A better understanding of the cognitive and functional impairments in schizophrenia-related conditions, as well as the identification of interventions that can reduce these impairments, are vital to improving outcomes for individual with these disorders.

DETAILED DESCRIPTION:
This study proposes to 1) evaluate the effects of 7.5 weeks of twice weekly cognitive remediation sessions, combined with concurrent administration of 8 weeks of guanfacine/placebo, on performance on cognitive, functional, and social skills performance measures in a sample of SPD patients with proven deficits in these areas. 2) Compare the effect of cognitive remediation therapy + 8 weeks guanfacine with cognitive remediation therapy + placebo on cognition in this schizophrenia spectrum disorder population. 3) Further characterize cognitive impairment in SPD using specific tests of working memory to evaluate the relationship between working memory and functional and social skill outcomes in this population.

The study hypothesizes that:

1. While both groups (those receiving CRT + guanfacine or CRT +placebo) will demonstrate improvements in overall cognitive functioning, SPD participants receiving CRT + guanfacine will evidence greater increases in post-treatment performance on our primary outcome measures-MATRICS battery total score, AX-CPT, N-Back, PASAT and DOT Test- particularly in areas related to working memory.
2. Participants receiving CRT + guanfacine will also demonstrate greater improvements in functional and social functioning exploratory measures, as evidenced by performance on our secondary assessments, the UPSA, SSPA, MASC, and Reading of the Mind in the Eyes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and having capacity to provide informed consent
* Currently meeting DSM-IV-TR criteria for Schizotypal Personality Disorder
* Males and females between the ages of 18-65
* Medically healthy: no major or partially treated medical condition that, based on the judgment of the clinician, would either put the patient at increased risk and/or affect our findings.
* Neurologically healthy: no brain injury or head trauma associated with loss of consciousness, seizures, or other conditions that may have caused functional impairment.
* At least two weeks free of medication while participating in this study
* Score at least one standard deviation below normative means on at least one test in the cognitive battery.
* At least 2 weeks free of psychotropic medication while participating in this study. Medication such as NSAIDS (e.g. Advil), Tylenol, Levothyroxine (if on stable dose 1 month, no symptoms of hypothyroidism and normal thyroid labs), non-centrally acting antihistamines, H2 blockers (e.g. Zantac), PPIs (e.g. Prilosec, Prevacid), and others that do not impact cognitive functioning will be allowed; the study physician will evaluate any medication at the time of the medical clearance on a case by case basis.

Exclusion Criteria:

* Meet criteria for bipolar I disorder, schizophrenia, schizoaffective disorder, or any other psychotic disorder Clinically significant cardiovascular or neurological conditions, uncontrolled hypertension, clinically significant EKG abnormalities, or serious general medial illness
* Current substance abuse or have met criteria for substance dependence within the last 6 months (excluding nicotine)
* Currently meeting DSM-IV-TR criteria for Major Depressive Disorder, not better accounted for and secondary to a personality disorder
* Currently taking psychotropic medications
* Currently taking any medications (systemic or otherwise) that the study physician determines could interfere with the study medication and put the participant at risk and/or interfere with the data
* Currently pregnant or lactating
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery Score | Baseline and 7.5 weeks after randomization
  Change in score at 7.5 weeks as compared to baseline. MATRICS Consensus Cognitive Battery: Subjects will complete the following MATRICS cognitive assessments. The dependent variable (DV) is the total MATRICS battery score. Trail Making Test (TMT): Part A Brief Assessment of Cognition in Schizophrenia: Symbol Coding (BACS SC) Hopkins Verbal Learning Test-Revised (HVLT-R) Weschler Memory Scale-III: Spatial Span Letter Number Span (LNS) Neuropsychological Assessment Battery (NAB): Mazes Brief Visuospatial Memory Test-Revised (BVMT-R) Category Fluency: Animal Naming

SECONDARY OUTCOMES:
Modified version of AX-Continuous Performance Test (AX-CPT) Score | Baseline and 7.5 weeks after randomization
  Change in score at 7.5 weeks as compared to baseline. This modified AX-CPT assesses context processing, a domain that has been shown to be impaired in both schizophrenia and SPD.
UCSD Performance Based Skills Assessment (UPSA) Score | Baseline and 7.5 weeks after randomization
  Change in score at 7.5 weeks as compared to baseline. The UPSA is an office based test to measure competence at performing day-to-day tasks in five domains: household chores, communication, finance, transportation, and planning recreational activities.
Social Skills Performance Assessment (SSPA) Score | Baseline and 7.5 weeks after randomization
  Change in score at 7.5 weeks as compared to baseline. The SSPA is an office based test designed to measure social competence.
Reading of the Mind in the Eyes Score | Baseline and 7.5 weeks after randomization
  Change in score at 7.5 weeks as compared to baseline. This is a measure of adult "mentalising", the ability to attribute mental states to oneself or another person.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNamara McClure, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] McClure MM, Barch DM, Romero MJ, Minzenberg MJ, Triebwasser J, Harvey PD, Siever LJ. The effects of guanfacine on context processing abnormalities in schizotypal personality disorder. Biol Psychiatry. 2007 May 15;61(10):1157-60. doi: 10.1016/j.biopsych.2006.06.034. Epub 2006 Sep 1. PMID 16950221
- [Background] Reichenberg A, Weiser M, Rapp MA, Rabinowitz J, Caspi A, Schmeidler J, Knobler HY, Lubin G, Nahon D, Harvey PD, Davidson M. Premorbid intra-individual variability in intellectual performance and risk for schizophrenia: a population-based study. Schizophr Res. 2006 Jul;85(1-3):49-57. doi: 10.1016/j.schres.2006.03.006. Epub 2006 Apr 19. PMID 16626941
- [Background] Heinrichs RW. The primacy of cognition in schizophrenia. Am Psychol. 2005 Apr;60(3):229-42. doi: 10.1037/0003-066X.60.3.229. PMID 15796677
- [Background] Friedman JI, Adler DN, Temporini HD, Kemether E, Harvey PD, White L, Parrella M, Davis KL. Guanfacine treatment of cognitive impairment in schizophrenia. Neuropsychopharmacology. 2001 Sep;25(3):402-9. doi: 10.1016/S0893-133X(01)00249-4. PMID 11522468
- [Background] Jakala P, Riekkinen M, Sirvio J, Koivisto E, Kejonen K, Vanhanen M, Riekkinen P Jr. Guanfacine, but not clonidine, improves planning and working memory performance in humans. Neuropsychopharmacology. 1999 May;20(5):460-70. doi: 10.1016/S0893-133X(98)00127-4. PMID 10192826